CLINICAL TRIAL: NCT02529683
Title: Clinical Trial of Acceptability, Adherence and Immune/Microbiologic Effects of a Vaginal Contraceptive Ring Among HIV-negative Women in Western Kenya
Brief Title: Study of Nuvaring Acceptability, Adherence and Biological Effects Among HIV-negative Women in Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Kenya Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CDC-NCHHSTP-6518; SSC Protocol # 2609 (Other: Kenya Medical Research Institute (FWA00002066))
Record Dates: First submitted 2015-08-14; First posted 2015-08-20 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Hormonal Contraception
Keywords: Nuvaring; contraceptive vaginal ring; Kenya; adherence; acceptability; immunological effects
MeSH Terms: interventions — NuvaRing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nuvaring (only arm) (Experimental): Nuvaring use for six months, with monthly pickup of rings and returning of used rings, and other behavioral/clinical assessments conducted during the visit on day 21 of the menstrual cycle.
  Interventions: Drug: Nuvaring

INTERVENTIONS:
Drug: Nuvaring — contraceptive vaginal ring with ethinyl estradiol and etonogestrel

SUMMARY:
One arm clinical trial of Nuvaring use for six months among 200 previously contracepting HIV-negative women (COCPs or DMPA) aged 18-35 in Kenya, where no vaginal rings are licensed/available for contraception or other indications. This was meant to be a formative research study to understand the predictors of acceptability and adherence to a contraceptive vaginal ring, and its immunoogical and microbiological effects over six months of product use.

DETAILED DESCRIPTION:
Background: Adherence to HIV prevention and contraception technologies is imperfect but a key to effectiveness. The options currently available to protect women from HIV infection and unwanted pregnancy (e. g. condom use, abstinence, monogamy) are not consistently available, practical, or under women's control. Intravaginal rings (IVRs) are an important technology that can be long-acting and woman-controlled and are being developed for HIV prevention with and without co-formulated hormonal contraception. Availability of IVRs in sub-Saharan Africa is limited; hence, it is important to evaluate acceptability, utilization, and biologic effects of IVR usage among African women. The NuvaRing® intravaginal combined hormonal contraceptive ring is used successfully in 61 countries worldwide, although not currently in Kenya. NuvaRing is self-inserted for 21 days starting after the last day of menses then removed for seven days to allow menses to occur, and has comparable effectiveness to oral contraceptives. Adherence to HIV prevention and contraception technologies like the IVR is critical to optimizing effectiveness. In preparation for a potential future Phase 2 trial of a combination antiretroviral-contraceptive IVR, KEMRI/CDC proposes to examine adherence, acceptability and biological effects of NuvaRing® among Kenyan women already using a modern method of contraception.

Objectives:

1. To assess adherence and utilization patterns for NuvaRing®, behaviourally and biologically.
2. To assess acceptability and effect of NuvaRing® on sexual behaviour among women and their sexual partners in a setting where there is no routine IVR use. At the end of the NuvaRing® trial, to additionally assess the hypothetical acceptability of a prototype dual use HIV-prevention and contraceptive IVR among women who had used NuvaRing® and among women who have never used an IVR.
3. To assess biologic effects of NuvaRing® including standard safety monitoring and, among a subset of participants, genital compartment immunology and microbiology.

Study Subjects: A total of 220 women and 20 men will be enrolled in different parts of the proposed study. The primary NuvaRing® trial participants (Objectives 1 and 2 above) will be up to 200 young, healthy women recruited from family planning clinics in the Kisumu catchment area. Fifty of these women will form a biomedical subgroup addressing Objective 3. To augment Objective 2, twenty trial participants and their sexual partners will take part in a qualitative in-depth interview, and three focus group discussions will be conducted, one with study participants and the others with 20 women who were not part of the primary NuvaRing® trial.

Design: Single arm clinical trial with up to 3 month pre-product phase (on oral or injectable contraceptives) followed by 6 months of IVR use, ending with an up to 3 month post-product phase during which women return to oral or injectable contraceptives and then exit the study. Monthly and quarterly follow-up will include adherence, acceptability and clinical assessments, and HIV and pregnancy testing. Women in the biomedical subgroup will undergo more frequent visits and collection of genital specimens. In-depth interview and focus group discussions are delineated under 'Study Subjects' above.

Outcome: The study will improve understanding of adherence to biomedical technologies, facilitate the conduct of future HIV microbicide clinical trials relying on IVR technology, and inform public health practice regarding contraception.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 34 years of age - Age will be verified using a standard national document e.g. Identity card, birth notification etc., and in case they are missing we will rely on proxy verification. Everyone in Kenya over the age of 18 is required to have a government-issued identification card, which includes their date of birth. There is some likelihood that women who are interested do not have this card and do not know their year of birth. In such, instances the participant will be asked her age and birth month. The day of birth will be defaulted to the 15th and year of birth will be calculated using the available information if not provided by the participant. In instances, where age cannot be verified, participation will not be permitted.
* Fluent in English, Swahili, or DhoLuo
* Resident of the Kisumu catchment area (≈150 kilometres from Kisumu City)
* Able and willing to provide written informed consent
* Willing to provide detailed locator information and not planning to relocate outside the study area for next 12 months
* Engaged in more than one episode of vaginal intercourse on different days in the past 30 days
* Female, not currently pregnant and not intending to get pregnant for the next 12 months
* Demonstrated willingness to prevent conception for the next 12 months, based on:

  o Documented receipt of three on-time monthly oral contraceptive pill (OCP) refills, or one DMPA injection at a FP clinic in the last 3 months prior to enrolling in the study.
* Willing to exclusively use IVR for contraception for the duration of the intervention phase of study. (Proper and consistent condom use will be encouraged and condoms will be provided for STI/HIV prevention)
* HIV negative per Kenya's HIV testing algorithm (using rapid tests)
* Willing to undergo periodic study procedures including pregnancy testing, HIV and STI testing

Exclusion Criteria:

* Participants will be excluded from the study based on:

  * Known medical contraindications:
  * Thrombophlebitis or thromboembolic disorders (current or history)
  * Cerebral vascular or coronary artery disease (current or history)
  * Valvular heart disease with thrombogenic complications
  * Severe hypertension
  * Diabetes with vascular involvement
  * Headaches with focal neurological symptoms
  * Major surgery with prolonged immobilization
  * Known or suspected carcinoma of the breast or personal history of breast cancer
  * Carcinoma of the endometrium or other known or suspected estrogen-dependent neoplasia
  * Undiagnosed abnormal genital bleeding
  * Cholestatic jaundice of pregnancy or jaundice with prior hormonal contraceptive use
  * Hepatic tumours (benign or malignant) or active liver disease
  * Known or suspected pregnancy
  * Heavy smoking (≥15 cigarettes per day) and over age 35
  * Hypersensitivity to any of the components of NuvaRing®
  * Current breastfeeding or being within three months of parturition, at the time of screening.
  * Evidence of clinically significant cardiac, respiratory, hepatic, gastrointestinal, endocrine, hematologic, psychiatric, neurologic, reproductive, or allergic disease that would compromise the ability of the participant to provide informed consent, or to complete study procedures or study requirements as determined by the principal investigator or designated associate. The clinical significance of any abnormality is to be evaluated in the context of the safety of the patient volunteer and the objectives of this study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2014-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Participant-reported Acceptability | Six months of product use
  Using computer assisted self-reported questionnaires and focus group discussions
Biological (Objective) measures of Adherence | Six months of product use
  Composite of salivary estradiol assays (instantaneous adherence) and remnant-drug assay of returned used vaginal rings (cumulative adherence over 21 days of use)
Local Immunological effects of vaginally delivered hormonal contraception as measured by immunophenotyping | Six months of product use
  Immunophenotyping analysis of cervicovaginal lavage collected at each day21 visit in a subset of participants, reported as total CD3, CD38 cell counts and proportions of CD4:CD8 cells
Participant-reported Adherence | Six months of product use
  Using computer assisted self-reported questionnaires and focus group discussions
Microbiological effect of vaginally delivered hormonal contraception | Six months of product use
  Standard Nugent score of cervicovaginal lavage smears.

CONTACTS AND LOCATIONS:
Overall Officials: Mumbi Makanga, MBChB, Study Chair — Kenya Medical Research Institute; Beatrice Nyagol, MN, Study Chair — Kenya Medical Research Institute; Eleanor McLellan-Lemal, PhD, Principal Investigator — US CDC; Mitesh Desai, MD, MPH, Study Chair — US CDC